CLINICAL TRIAL: NCT00065286
Title: Movement Dynamic Analyses of Akathisia
Brief Title: Akathisia (Restless Legs Syndrome) in People With Schizophrenia and Mental Retardation
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: 5R01HD034027 (NIH); NICHD-17; 5R01HD034027 (NIH)
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Akathisia
Keywords: Akathisia; Mental retardation; Schizophrenia; Neuroleptic medication; Tardive dyskinesia; Brief Psychiatric Rating Scale; Barnes test; Stereotypy Checklist Test; DISCUS Tardive Dyskinesia test
MeSH Terms: conditions — Psychomotor Agitation; Intellectual Disability; Schizophrenia; Tardive Dyskinesia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Akathisia is a movement disorder that is often a side effect of certain psychiatric drugs. People with akathisia are unable to sit or keep still, complain of restlessness, fidget, rock from foot to foot, and pace. Akathisia is sometimes called "restless legs syndrome." The drugs that can cause akathisia are most often used to treat patients with schizophrenia or mental retardation (MR). This study will evaluate akathisia in both schizophrenic and MR patients who either have long-term akathisia or who are starting treatment with psychiatric drugs.

DETAILED DESCRIPTION:
Akathisia is a relatively common side effect of neuroleptic medication that occurs within 1 week to 6 months after the initiation of medication. Akathisia is characterized by a variety of movement manifestations, such as fidgeting, irritability, inability to sit or stand still, marching in place, continuous trunk motions, sleeplessness, and a subjective sense of restlessness. Akathisia has been studied primarily in schizophrenic patients, although reports on individuals with mental retardation suggest that akathisia also occurs in this population. This study will characterize the movement dynamics of akathisia in schizophrenic and mentally retarded adults using two experimental series.

The first experimental series will compare chronic akathisia in schizophrenic and MR patients. Four groups of MR patients and four groups of schizophrenic patients will be studied: young (age 18 to 38) with chronic akathisia, older (age 40 to 60) with chronic akathisia, young on neuroleptics without akathisia, and older on neuroleptics without akathisia. Two control groups will include healthy individuals with normal intelligence who are not on neuroleptic medication. Assessments will include videotaped recordings and kinematic analysis of naturally occurring akathisia restlessness movements as well as cognitive and psychiatric tests. Demographic factors (age and sex) and medication factors (type and duration) will also be assessed to determine their relation to and possible impact on chronic akathisia.

The second experimental series will compare schizophrenic and MR patients who are initiating neuroleptic therapy. Institutionalized MR patients will be age matched with schizophrenic patients. Tests will occur at baseline (prior to drug initiation) and at Weeks 1, 2, 4, 8, 16, 24, and 52. Those who enroll in the protocol early will be tested for more than 12 months where possible and useful. The same analyses as in the first experimental series will be used to allow for comparison of acute and chronic akathisia.

ELIGIBILITY:
Inclusion Criteria for Experimental Series I

* Chronic akathisia for at least 3 months prior to study entry
* Neuroleptic medication for at least 6 months prior to study entry (anticonvulsant medication will be accepted and those on carbamazepine and ethosuximide will be monitored for the development of akathisia)
* Mental retardation/developmental delay diagnosis based on American Association of Mental Deficiency definition or diagnosis of schizophrenia based on the DSM-IV criteria

Inclusion Criteria for Control Group

* Control groups will be matched to akathisia groups based on age and level of disability (IQ for mental retardation population, BPRS positive symptoms of schizophrenia for schizophrenic groups).

Exclusion Criteria

* Psychotropic drugs such as serotonin re-uptake inhibiting anti-depressants
* Nonambulatory
* Uncontrolled seizure disorders
* Fragile X syndrome
* Down Syndrome
* Neurological disease that is known to have definitive symptoms of choreoathetosis, dystonia, Syndenham's chorea, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 1996-12; Study Completion 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Karl M Newell, Ph. D., Principal Investigator — Department of Kinesiology
Locations (2):
- United States (2):
  - Western Carolina Center, Morganton, North Carolina
  - Department of Kinesiology, University Park, Pennsylvania

REFERENCES:
- [Background] Newell KM, Incledon T, Bodfish JW, Sprague RL. Variability of stereotypic body-rocking in adults with mental retardation. Am J Ment Retard. 1999 May;104(3):279-88. doi: 10.1352/0895-8017(1999)1042.0.CO;2. PMID 10349469
- [Background] Newell KM, Bodfish JW, Mahorney SL, Sprague RL. Dynamics of lip dyskinesia associated with neuroleptic withdrawal. Am J Ment Retard. 2000 Jul;105(4):260-8. doi: 10.1352/0895-8017(2000)1052.0.CO;2. PMID 10934568
- [Background] Newell KM, Wszola B, Sprague RL, Mahorney SL, Bodfish JW. The changing effector pattern of tardive dyskinesia during the course of neuroleptic withdrawal. Exp Clin Psychopharmacol. 2001 Aug;9(3):262-8. doi: 10.1037//1064-1297.9.3.262. PMID 11534536
- [Background] Newell KM, Ko YG, Sprague RL, Mahorney SL, Bodfish JW. Onset of dyskinesia and changes in postural task performance during the course of neuroleptic withdrawal. Am J Ment Retard. 2002 Jul;107(4):270-7. doi: 10.1352/0895-8017(2002)1072.0.CO;2. PMID 12069646